CLINICAL TRIAL: NCT06917027
Title: Comparison of Mobile Education and Face-to-Face Intermittent Catheterization Education in Terms of Knowledge and Skill Levels of Nursing Students
Brief Title: Comparison of Mobile Education and Face-to-Face Intermittent Catheterization Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nilgün Aras, PhD, nurse, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E.1200559
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Neurogenic Bladder
Keywords: neurogenic bladder; intermittent catheterization; education; nursing student
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: parallel group, randomized, controlled trial
Masking Description: Blocked randomization was used for the groupings by a person independent of the researchers using a computer random-sequence generator (http://randomizer.org).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (face to face education) (Other): Students in the face-to-face education group will receive theoretical training on intermittent catheterization. In addition, the CIC procedure steps will be explained with a demonstration technique. One week after the face-to-face education group is trained, the participants will perform intermittent catheterization in the laboratory and complete the final tests.
  Interventions: Other: education
- experimental group (education with mobil application) (Experimental): On the day the face-to-face education group is trained, the mobile application will be loaded onto the mobile education group phones. The videos in the mobile application will be introduced to the participants and made available for use. One week after the mobile application is loaded onto the mobile education group, the participants will perform intermittent catheterization in the laboratory and complete the final tests.
  Interventions: Other: education

INTERVENTIONS:
Other: education — clean intermittent catheterization education

SUMMARY:
Today, Clean Intermittent Catheterization (CIC) is widely used to drain urine accumulated in the bladder in acute or chronic problems such as neurogenic bladder and prostate hypertrophy.The success of the technique depends largely on patient education and follow-up.Nurses play a fundamental role in providing theoretical and practical learning in CIC training and early detection of complications. Although face-to-face education is widely used in the education of nursing students, mobile applications have become popular in recent years. There is no previous study in the literature on clean intermittent catheterization education with nursing students. The purpose of this study is to compare mobile-assisted education with face-to-face intermittent catheterization education in terms of knowledge and skill levels of nursing students.

DETAILED DESCRIPTION:
Today, Clean Intermittent Catheterization (CIC) is widely used to drain urine accumulated in the bladder in acute or chronic problems such as neurogenic bladder and prostate hypertrophy.Since CIC is a procedure performed on the bladder, it may cause some complications.In order to prevent or reduce complications, CIC application must be performed successfully. The success of the technique depends largely on patient education and follow-up.Nurses play a fundamental role in providing theoretical and practical learning in CIC training and early detection of complications.For this reason, it is important for nurses to have knowledge on this subject in terms of the quality of the education to be given and patient follow-up. Although there are international guidelines in the literature prepared for nurses who will provide CIC training, nursing students' knowledge on this subject is generally limited to indwelling urinary catheterization.Today, the rapid development of technology and pandemics such as COVID-19 have shown the importance of alternative education methods in addition to face-to-face education. Educational technologies are used in nursing education and these methods provide student-centered education to students wherever and whenever they want.It is important for nursing students to understand this issue better through mobile applications and face-to-face training, and to know how to communicate with the patient and what materials will be needed when a patient who applies CIC is admitted to the hospital. Because although CIC training is given by professional nurses in urology and rehabilitation clinics, patients who apply CIC may be admitted to different clinics due to other health problems. In such cases, the nurse working in the clinic must have knowledge about CIC application. Although face-to-face education is widely used in the education of nursing students, mobile applications have become popular in recent years. There is no previous study in the literature on clean intermittent catheterization education with nursing students. The purpose of this study is to compare mobile-assisted education with face-to-face intermittent catheterization education in terms of knowledge and skill levels of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student,
* Being willing to participate in the research,

Exclusion Criteria:

* The student in the mobile-assisted education group did not watch the videos in the mobile application,
* The student in the face-to-face education group did not attend the training,
* The student did not complete the pre-test or post-test/completed it incompletely,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
"intermittent catheterization check-lists" | The checklists were filled out by the researchers 7 days after the training, based on the participants' implementation success.
  Intermittent catheterization check-lists evaluates the clean intermittent catheterization procedure steps. The female checklist consists of 21 items, the male checklist consists of 23 items. Each correct answer is worth 1 point, and each wrong/incomplete answer is worth 0 points. The female checklist has a maximum of 21 points, and the male checklist has a maximum of 23 points.
  The checklists were filled out by the researchers 7 days after the training, based on the participants' implementation success.
clean intermittent catheterization knowledge form | The knowledge form was filled out by the participants 7 days after the training.
  The knowledge form aims to evaluate the participants' knowledge of clean intermittent catheterization. It consists of 17 questions. A minimum of 0 - a maximum of 17 points can be obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared with other researchers.